CLINICAL TRIAL: NCT06226337
Title: The Effect of Music on Pain and Anxiety During Hysterosalpingography: A Randomised Controlled Trial
Brief Title: The Effect of Music on Pain and Anxiety During Hysterosalpingography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ayse Aydin, Dr. Lecturer, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BMumcu
Record Dates: First submitted 2024-01-04; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Hysterosalpingography
Keywords: hysterosalpingography; nursing; pain; anxiety; music
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention: control group (No Intervention): No intervention was applied to the control group other than routine practice.45 women were assigned to the control group
- Experimental group (Experimental): 45 women to the experimental group. In the study, the experimental group Acemaşiran makam was played to the women as music during hysterosalpingography.
  Interventions: Other: listen music

INTERVENTIONS:
Other: listen music — During hysterosalpingography, women were listened to the Acemaşiran maqam as music via MP4 players and headphones.
  Arms: Experimental group

SUMMARY:
This randomised controlled experimental study was conducted at the Gynecology Polyclinic of Atatürk University Health Research and Application Center between 27.01. 2022 and 04.12.2023. Population of the study consisted of women admitted to the relevant institution for hysterosalpingography.

Sample of the study consisted of a total of 80 women, 40 in the experimental group and 40 in the control group, who met the research criteria from the specified population. In the study, the women in the experimental group were listened to Acemaşiran makam as music during hysterosalpingography. No intervention was applied to the control group except routine practice. "Personal Information Form", "Visual Analogue Scale (VAS)" and "State Anxiety Scale" were used to collect the data.

DETAILED DESCRIPTION:
Hysterosalpingography (HSG) is a diagnostic radiological procedure used widely to investigate infertility as an invasive, uncomfortable, and painful procedure. The purpose of the present study was to examine the effects of music played to women during Hysterosalpingography on pain and anxiety.

Study design: The study had a randomized-controlled double-blind design. Setting and Sample: The population of the study consisted of women who applied to the Gynecology outpatient clinic of Atatürk University Health Study and Application Center between 01.06.2023 and 01.11.2023 to undergo Hysterosalpingography. HSG scans are performed in the Radiology Unit of the hospital. The sample number of the study was calculated by using the G*Power Program (version 3.1.9.6). The number of samples for each group was calculated as 35 in the calculation, with a large effect size (d = 0.80), 5% margin of error (α = 0.05), and 95% power (1-β = 0.80). Considering the possibility of data losses, the number of samples was increased by 10 for each group and it was planned to include 45 participants in each group (a total of 90 people in the sample). A total of 45 women were assigned to the Experimental Group and 45 women to the Control Group with the Simple Randomization Technique. Five people from the Control Group (they did not fill out the post-test data collection tool) and five people from the Experimental Group (three people left at their own request, and two people were excluded because they used analgesics) were excluded from the study during the study period. The study was completed with 80 women (40 in the Experimental Group and 40 in the Control Group).

Inclusion and Exclusion Criteria Inclusion criteria Being over 18 years of age, being at least a primary school graduate, agreeing to participate in the study voluntarily, having no active infections, no vaginal bleeding on the day of the procedure, not having had an HSG before, not receiving sedation, not having a hearing problem, and not having any obstacle to wearing headphones (for the Experimental Group), not taking any medications that might affect blood pressure and pulse rate (e.g., Digoxin, Adrenaline), and not having a diagnosed psychiatric disease.

Exclusion Criteria Using analgesics before or after the procedure, using antidepressants or sedative medications, being allergic to radio-opaque material, not completing the procedure, not completing one of the pre-test or post-test forms, filling in incomplete data, and leaving the study voluntarily.

Data Collection and Procedure Data Collection The data of the study were collected with the face-to-face interview technique between 01.06.2023 and 01.11.2023 by a neutral researcher (a nurse) who was not familiar with the groups trained by the researcher. The women participating in the study were interviewed at the clinic where they applied for the procedure, the purpose and stages of the study were explained, and they were told that they could withdraw at any stage of the study. Before starting to collect the study data, women were informed about the study, and their consent was obtained. It took an average of 5-10 minutes for each patient to fill out the forms.

Hysterosalpingography Procedure HSG is performed three days a week (Monday, Wednesday, and Thursday) in the Radiology Unit after the decision of the gynecologist. The patient makes an appointment for an HSG examination at the gynecology clinic, based on the last menstrual date. The patient comes to the polyclinic and gives blood to rule out pregnancy on the morning of the HSG scan. At 13:00, she is taken to the Radiology Unit for an HSG scan. The procedure is performed in the lithotomy position. A water-soluble contrast agent (KOPAQ-350 mgl/ml) is injected slowly. Fluoroscopic images are taken intermittently to evaluate the uterus and fallopian tubes. After the HSG procedure, the result is evaluated by the physician.

Nursing Intervention Used in the Study: Music Expert opinion was taken from the Turkish Music Research and Application Center (TUMATA) in determining the music that would be played to the patients. The Maqam that TUMATA recommended for this study was "Acemaşiran Maqam". Acemaşiran Maqam was used in the study because of its pain-relieving and spasm-relieving characteristics and its ability to promote relaxation. The women in the Experimental Group were allowed to listen to music for an average of 15 minutes during the HSG procedure as a nursing intervention. When the patient was laid on the table for the procedure, she was given headphones, and music was played on the MP4 player. HSG lasted approximately 15 minutes. Each patient was given disposable headphones because of hygiene conditions.

Control Group A personal information form was used 10 minutes before the HSG procedure. The patients were asked to fill out the State Anxiety Inventory to determine their anxiety level as a pre-test. Pain was not measured before the procedure because pain develops in women because of the HSG procedure. The women were told that they would be asked to refill the relevant measurement tools for the post-test after the procedure, they were told to write a nickname that would be easy to remember later in the nickname section of the form, and the "Visual Analog Scale" and the "State Anxiety Inventory" were filled in as the post-test 10 minutes after the procedure.

Human Subjects Protection Approval was obtained from Atatürk University Faculty of Medicine Clinical Study Ethics Committee before starting the study (27/01/2022 with the decision number 1/16). Written permission was obtained from the institution where the study was conducted (21/11/2022 with the number 2200382092). The patients were informed about the study and their consent was obtained before starting to collect study data. It was also stated that personal information would not be disclosed to third parties through an "Informed Consent Form" and that care would be taken to comply with the "Principle of Confidentiality and Protection of Confidentiality". The "Anonymity and Security principle" was fulfilled by keeping the data and the identity of the participant confidential. The Principles of the Declaration of Helsinki were followed throughout the study.

Statistical Analysis The data were evaluated in the Statistical Package for the Social Sciences (SPSS) 22 package program. The data were analyzed for normality by using kurtosis and skewness. The threshold for statistical significance was taken as p < 0.05.

ELIGIBILITY:
Inclusion criteria Being over 18 years of age, being at least a primary school graduate, agreeing to participate in the study voluntarily, having no active infections, no vaginal bleeding on the day of the procedure, not having had an HSG before, not receiving sedation, not having a hearing problem, and not having any obstacle to wearing headphones (for the Experimental Group), not taking any medications that might affect blood pressure and pulse rate (e.g., Digoxin, Adrenaline), and not having a diagnosed psychiatric disease.

Exclusion Criteria Using analgesics before or after the procedure, using antidepressants or sedative medications, being allergic to radio-opaque material, not completing the procedure, not completing one of the pre-test or post-test forms, filling in incomplete data, and leaving the study voluntarily.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Have Hsg done
Enrollment: 80 (Actual)
Dates: Start 2022-01-22 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | 5 months
  Personal Information Form:The form, which was prepared by the researcher in line with the literature data, included 10 questions
State Anxiety Inventory | 5 months
  There are 20 questions in the state part of the scale providing a four-point Likert-type measurement. On the scale, the scoring varies between 1 (not at all) and 4 (completely). One point indicates that the situation stated in the question does not reflect the individual at all, and 4 points indicate that the situation reflects the individual completely. The highest score is 80 and the lowest score is 20. A high total score indicates that the individual's anxiety level is also high.The scores between 20 and 37 indicate no or minimal anxiety, scores between 38 and 44 indicate moderate anxiety, and scores between 45 and 80 indicate high anxiety on the State Anxiety Inventory.
Visual Analog Scale (VAS) | 5 months
  Visual Analog Scale is an evaluation tool in which patients mark on a 10 cm ruler. The 10 cm scale, which is a numerical pain assessment scale, starts with "No pain (0)" and ends with "Unbearable pain (10)". The patient is asked to mark the place that expresses his/her pain on the line. The distance marked by the patient is measured by taking the zero starting distance. The pain level of the patient is determined in this way. The horizontally prepared VAS was used to evaluate pain intensity in this study. The reason for choosing this scale in the study was that it is easily understandable by the participants and easy to use.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe AYDIN, Dr. Lecturer, Study Director — Ataturk University Faculty of Nursing
Locations (1):
- Ataturk University Faculty of Nursing, Erzurum, Yakuti̇ye, Turkey (Türkiye)